CLINICAL TRIAL: NCT06605443
Title: Precision Medicine for L/GCMN and Melanoma 1 (Precis-mel 2)
Brief Title: Precision Medicine for L/GCMN and Melanoma 2
Acronym: Precis-mel 2
Status: Recruiting | Type: Observational
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2023/1111; HORIZON-MISS-2021-CANCER-02-03 (Other Grant/Funding Number: European Comission)
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-09

CONDITIONS: Melanoma (Skin Cancer); Nevi and Melanomas; Congenital Melanocytic Nevus
Keywords: Volatilomics; Breath analyzer; Skin patch; Melanoma; L/GCMN; Liquid biopsy; cfDNA; Non-invasive diagnostics
MeSH Terms: conditions — Melanoma; Nevi and Melanomas | interventions — Transdermal Patch; Liquid Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell-free DNA will be extracted from patient blood and saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Melanoma (non-metastatic): Patients of either sex over 18 years old with histopathological confirmed melanoma in a non metastatic stage (I to IIb stages according to AJCC classification)
  Interventions: Device: Breath analyzer; Device: Skin patch; Genetic: Liquid biopsy
- Melanoma (metastatic): Patients of either sex over 18 years old with histopathological confirmed melanoma in a metastatic stage (IIIa to IV stages according to AJCC classification)

INTERVENTIONS:
Device: Breath analyzer — The study subject will be advised to sit quietly for minimum 10 minutes prior the sampling to avoid temporal changes in levels of volatile organic compunds (VOCs) related to body movement or try to avoid abrupt changes in body posture. Then, he/she will be asked to blow in the breath analyzer in order to obtain the exhaled VOCs profile.
  Groups: Melanoma (non-metastatic)
Device: Skin patch — A skin patch will be placed in the anterior part of the patient's arm for the obtention of the skin VOCs profile (estimated sampling time of around 1 h). These profiles will be recorded with a dedicated software and analyzed using standard statistical methods.
  Groups: Melanoma (non-metastatic)
Genetic: Liquid biopsy — Circulating free tumor DNA (cfDNA) will be extracted from patient's blood and analyzed to detect mutations in BRAF and other prognostic genes.
  Groups: Melanoma (non-metastatic)

SUMMARY:
The primary objective is to evaluate the possibility of using minimally and non-invasive technologies (skin patch and breath analyzer) based on the detection of volatile organic compounds (VOCs) for the early identification of metastases. The secondary objective is to evaluate the usability of these technologies in the follow up of high-risk melanoma patients.

DETAILED DESCRIPTION:
This is a unicentric national prospective observational study aimed at evaluating the use of two devices (skin patch and breath analyzer) for the non or minimally invasive diagnosis of metastatic melanoma with a total duration of 24 months. The study will be based on the obtention of different patterns of volatile organic compounds using the aforementioned devices for melanoma patients with and without metastasis. The results will be compared with the standard procedures for the detection of metastatic melanoma (standard imaging techniques such as PET, MRI, etc.) and correlated with standard prognostic biomarkers (cfDNA mutations in BRAF, NRAS, etc.) obtained using liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Have a histopathological confirmed melanoma diagnosis (stage II, III or IV AJCC)

Exclusion Criteria:

* Not signing the informed consent form
* Present other cancers or chronic diseases (such as diabetes, asthma, etc.), which may affect the volatile organic compound profiles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population (over 18 years of age) diagnosed with melanoma that are currently being treated at the Hospital Clinic de Barcelona or that are admitted before or at the time of the enrolment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Early identification of metastases | 24 months
  The primary objective of the study is to evaluate the possibility of using minimally and non-invasive technologies (skin patch and breath analyzer) based on the detection of volatile organic compounds (VOCs) for the early identification of metastases.

SECONDARY OUTCOMES:
Follow-up of high-risk melanoma patients | 24 months
  The secondary objective is to evaluate the possibility to follow-up high risk melanoma patients using minimally invasive technologies based on the detection of changes in the patterns of volatile organic compounds (VOCs).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Clínic de Barcelona (Dermatology service), Barcelona
  - Hospital Clínic Barcelona, Barcelona